CLINICAL TRIAL: NCT03849352
Title: Can People Living With and Beyond Colorectal Cancer Make Lifestyle Changes With the Support of Health Technology
Brief Title: Lifestyle Changes Using Digital Technology in Colorectal Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CCR5040
Record Dates: First submitted 2019-02-18; First posted 2019-02-21 (Actual); Last update posted 2019-02-21 (Actual); Status verified 2019-02

CONDITIONS: Life Style; Colo-rectal Cancer
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lifestyle Arm (Other): Can people living with and beyond colorectal cancer make lifestyle changes with the support of health technology
  Interventions: Behavioral: Lifestyle changes with the support of health technology

INTERVENTIONS:
Behavioral: Lifestyle changes with the support of health technology — Written instructions will be provided to participants, to include how to download supportive apps on smartphones. Participants will be asked to complete a 3 day food diary using an online platform (MyFood24) prior to attending a face to face consultation which will reinforce the participant's responsibilities. Participants will be assisted to set specific diet and lifestyle goals. 3 fortnightly follow ups will be arranged via 15 minute telephone consultations, three 24 hour dietary diaries will be completed via MyFood24 prior to each fortnightly digital consultation. Participants will be asked to measure their daily activity via a pedometer on their smart phones. Participants will be asked to complete the Godin leisure time questionnaire to assess changes in leisure time exercise.

SUMMARY:
The objective of this small study is to assess the feasibility of remotely delivering a diet and lifestyle intervention following treatment of CRC through telecommunications and digital technology. A DBCI will be implemented among a population of people living with and beyond CRC to help identify if patients find this an easy and achievable way to communicate with a Registered Dietitian. The information gained from this small scale feasibility will be used to help develop a larger study on supporting people with CRC to make a lifestyle change.

DETAILED DESCRIPTION:
Fifty four percent of Colorectal cancer (CRC) cases are thought to be preventable, showing it has a strong correlation with lifestyle factors. A recent report by the World Cancer Research Fund and American Institute of Cancer Research (WCRF/AICR) on diet, physical activity (PA) and CRC reported numerous findings linking lifestyle with primary prevention of CRC. Approximately six out of ten people diagnosed with bowel cancer in England and Wales survive for 10-years or more and rates of survival have more than doubled in the last 40-years.

The term 'cancer survivors' denotes all people who are living with a diagnosis of cancer, and those who have recovered from the disease. The term is not universally accepted and survivors are increasingly being referred to as people 'living with and beyond cancer. This covers a wide variety of circumstances including people at diagnosis, during and post treatment, and those with recurrence therefore including people with potentially differing nutritional needs. People can be struggling with a poor nutritional intake due to treatment side effects or may need to optimise their nutritional status preoperatively or require advice post treatment for optimum recovery and rehabilitation. However, compared to the vast amount of research with respect to CRC incidence there is a paucity of research on diet and lifestyle factors influencing CRC recurrence and survival.

The second WCRF and AICR expert report in 2007 undertook a systematic literature review to assess the role of food, nutrition and PA in people diagnosed with cancer. The report included randomized control trials (RCTs) evaluating dietary interventions, however, there were no conclusions drawn. This was attributed to poor quality designs and varying intervention duration of the studies. The third WCRF and AICR expert report, in 2018, stated new evidence had accrued since the second report but primarily within breast cancer therefore a review of the evidence was undertaken in this group leaving a gap in the evidence base with regard to CRC.

The design of secondary prevention studies are based on expert conclusion with the third WCRF recommending survivors who have completed treatment should follow the general advice for cancer prevention. The current strongest primary prevention evidence is that CRC risk is decreased by being physically active in addition to a higher consumption of wholegrains, dietary fibre and dairy products. Risk is increased by the consumption of red and processed meat, more than two alcoholic drinks per day and being overweight or obese.

A recent review of the literature of lifestyle interventions in RCTs in people with CRC has identified 6 published studies (in preparation). The review identified that all current studies used a variety of dietary and physical activity interventions, data collection tools and inconsistent timing of interventions commencing from 6 months to 5 years post diagnosis. None of the published RCTs achieved changes in dietary intake and any small changes that occurred were not sustainable with participants reverting to their usual dietary habits.

One conclusion from the review was that no studies used appropriate methods to support behaviour change such as healthcare professionals trained in behaviour change techniques and methods of support, for example, digital technology. It has been demonstrated that such techniques would help support people to make lifestyle changes and from a research perspective can eliminate administration-intensive tasks, variation in interpretation and recording errors

Discussion with the PPI group of The Royal Marsden Hospital (NHS Foundation Trust) and Institute of Cancer Research provided a valuable insight into the variance in opinion as to when and how people could be asked to make lifestyle changes. The support provided by family members and / or carers was identified as a critical factor in supporting people to make lifestyle changes.

There has recently been an increased interest in the use of digital behaviour change interventions (DBCIs) and smartphone applications in the healthcare setting, including in the management of diet, PA and weight.

A recent systematic review of DBCIs amongst cancer survivors identified fifteen studies and concluded DBCIs can improve PA and Body Mass Index (BMI), in this patient group, with mixed results for improved dietary behaviours.

ELIGIBILITY:
Inclusion Criteria:

1. All adult outpatients, over the age of 18, under The Royal Marsden NHS Foundation Trust with a formal diagnosis of stage I-III CRC.
2. Participants must have completed treatment for CRC (defined as 3 weeks after stopping chemotherapy) and own a smart phone.

Exclusion Criteria:

1. Patients who have metastatic disease
2. Patients who have experienced a significant weight loss >10% body weight in past 3 months as they are at risk of malnutrition and will be referred to the dietitians for advice beyond healthy living and diet advice.
3. Patients with a BMI >35 kg/m2
4. People with a prior formal diagnosis of memory impairment
5. Patients who cannot read or write English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-03-18 (Estimated); Primary Completion 2019-05-03 (Estimated); Study Completion 2019-06-14 (Estimated)

PRIMARY OUTCOMES:
To evaluate whether patients who have undergone CRC treatment are able to comply with remote follow-ups using telephone reviews and digital technology to help promote and track individual healthy lifestyle, diet and PA changes. | Week 2 after patient recruitment
  Mean percentage of CRC patients who have been able to engage with remote reviews through telecommunications and digital technology at the end of the 2 month intervention. This will be defined as patients that either have completed an online food diary or engaged with the dietitian over the telephone to set and monitor their diet and lifestyle changes.

SECONDARY OUTCOMES:
To examine the demographics of people with CRC who are willing to participate in a study focused on lifestyle changes | Week 1 after patient recruitment
  The demographics including but not limited to age and gender of patients
To ascertain the proportion of CRC patients willing to interact with the intervention | Week 5 after patient recruitment
  Proportion of patients willing to take part in this study. This will be defined as those accepting to register to the study by completing the baseline three day food diary out of those approached to take part.
To identify participant reported barriers and acceptability of the use of remote reviews using telephones and digital technology | study completion
  Specific barriers preventing the remote follow ups using telecommunications and digital technology for diet and lifestyle changes will be identified and their frequency and percentages will be reported. These will be recorded on an end of intervention evaluation form and the analysis will be mainly qualitative.
To explore the frequency of telephone contact by participants during the 2 month intervention | Week 10 after patient recruitment
  The number and duration of telephone calls between dietitian and participant will also be summarized.
To explore how much time is required for a healthcare professional to deliver the healthy diet and lifestyle intervention | Study completion
  Measure how much time is required to deliver the intervention by dietitians. The dietitian will log on a spread sheet time spent arranging appointments and interacting with participants in person and the telephone
To ascertain whether there was any change in diet and lifestyle factors from baseline to end of intervention (2 months) | Study completion
  The proportion of participants that had a change in their diet (defined as increased fibre and fruit and vegetables, decreased red meat, processed meat and alcohol) as assessed by comparing parameters from the baseline and end of intervention (at 2 months) three day food diary

CONTACTS AND LOCATIONS:
Overall Officials: Clare Shaw, BSc, PhD, Principal Investigator — Royal Marsden NHS Foundation Trust

REFERENCES:
- [Derived] Nelson V, Cross AJ, Powell J, Shaw C. Can people living with and beyond colorectal cancer make lifestyle changes with the support of health technology: A feasibility study. J Hum Nutr Diet. 2023 Apr;36(2):554-565. doi: 10.1111/jhn.13008. Epub 2022 Apr 9. PMID 35320595